CLINICAL TRIAL: NCT06055647
Title: Evaluation of Immunohistochemical Expression of Human Epidermal Growth Factor Receptor 2 (HER 2) and Its Association With Clinicopathological Variables in Patients With Pancreatic Duct Adenocarcinoma in Upper Egypt
Brief Title: HER-2 Expression in Pancreatic Duct Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Maisa Hashem Mohammed, Maisa H Mohammed, MD, Sohag University
Other Study IDs: Soh-Med-23-09-4PD
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: HER-2; Pancreatic Duct Adenocarcinoma; Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: immunohistochemical approach — Formalin-fixed, Paraffin-embedded tissue blocks of pancreatic duct adenocarcinoma will be stained by anti HER-2, by immunohistochemical approach.

SUMMARY:
Pancreatic duct adenocarcinoma is a highly aggressive carcinoma that is associated with a poor prognosis. Detection of novel biological markers that are specifically over expressed in pancreatic duct adenocarcinoma and their subsequent targeting by anti cancer therapeutic modalities may improve patient's survival.

DETAILED DESCRIPTION:
Pancreatic duct adenocarcinoma (PDAC) is a deadly neoplasm that showed current increase in its occurrence. There are many challenges in PDAC; the tumor is frequently associated with perineural invasion and angioinvasion, these lead to early metastasis.Another important challenge is that the tumor is associated with extensive fibrosis that prevents arrival of chemotherapeutic agents. Most modern anti-cancer therapeutic modalities depend on the biologic signature of the tumor. Human epidermal growth factor receptor-2 (HER-2) is a cell surface protein that is associated with enhanced cellular proliferation. HER-2 has been detected and successfully targeted in many human carcinomas as breast and gastric cancers. we aimed to evaluate the potential cancer-promoting effect of HER-2 in PDAC, in order to detect any possible benefits of its targeting by future therapeutic modalities.

ELIGIBILITY:
Inclusion Criteria:

1. Cases of PDAC who underwent radical operations.
2. Tissue blocks with sufficient material.
3. Cases with available clinical data.

Exclusion Criteria:

1. Cases of pancreatic carcinoma other than PDAC.
2. Patients who received preoperative chemotherapy or radiotherapy.
3. Patients with PDAC who were diagnosed by tru-cut biopsies only and didn't undergo radical operations.
4. Cases with insufficient/destructed material.
5. Patients with inadequate clinical data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: • This study will be performed on archived formalin-fixed, paraffin-embedded tissue blocks that belonged to 37 patients who were admitted to Assuit and Sohag Oncology Centers and Sohag university hospital from January, 1st, 2017 to December, 31st, 2020. Patients' complaints included obstructive jaundice, abdominal pain and vomiting. Radiological assessment revealed heterogeneous suspicious pancreatic lesions from which tru-cut biopsies were obtained and examined by the standard staining method; hematoxylin and eosin (H&E). Cases diagnosed as pancreatic carcinoma on the basis of tru-cut biopsies underwent pancreaticoduodenectomy (Whipple procedure) or distal pancreatectomy, depending on tumor location.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
correlation of HRE-2 expression with clinical and pathological parameters | 6 months
  levels of HER-2 expression will be correlated with clinical parameters (as patients' ages, sexes, tumor location), and pathological parameters (as tumor grades, stages, neural and vascular invasion).

IPD SHARING:
Plan to Share IPD: Undecided